CLINICAL TRIAL: NCT04498416
Title: Methodology of " CoCo 20 ": a Longitudinal Follow-up Study of the Paediatric Population and Their Families During and After the Coronavirus Pandemic and the Confinement
Brief Title: CoCo-20: a Longitudinal Follow-up Study of the French Paediatric Population During and After the Coronavirus Pandemic COVID-19
Acronym: CoCo-20
Status: Completed | Type: Observational
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Other Study IDs: 20-HPNCL-05
Record Dates: First submitted 2020-07-31; First posted 2020-08-04 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-01

CONDITIONS: Mental Health Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 Post-Traumatic Stress Disorder (PTSD): children with an identified traumatic history
  Interventions: Diagnostic Test: Quantitative and qualitative assessments of mental health
- Group 2 Pathology: children with psychological follow-up treatment for a psychiatric disorder, without traumatic history;
  Interventions: Diagnostic Test: Quantitative and qualitative assessments of mental health
- Group 3 Control: children without traumatic experience and without psychiatric or psychological follow-up treatment.
  Interventions: Diagnostic Test: Quantitative and qualitative assessments of mental health

INTERVENTIONS:
Diagnostic Test: Quantitative and qualitative assessments of mental health — Emergency semi-directed interview; Diagnosis Infant and Preschool Assessment (DIPA); Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS); Conners Scale - short version;Weiss functional impairment rating scale - parent (WFIRS); Parenting stress index-short form (PSI-SF); Anxiety Scale

SUMMARY:
In the context of a viral outbreak and of widespread quarantine measures, a significant increase in psychological disorders, such as stress or fear behaviours, had previously been observed. This distress has been described on adults, but no data have been collected yet for paediatric populations.

After a traumatic event, children and adolescents may present several clinical consequences, the most common being Post-Traumatic Stress Disorder (PTSD). Moreover, PTSD in children and adolescents is often associated with comorbid disorders, such Attention Deficit Hyperactivity Disorder, depression, attachment and anxiety disorders, sleep disturbances and behavior problems.

The aim of this study is to present the methodology of "CoCo 20" : is to assess the impact of the pandemic of coronavirus disease 2019 (Covid-19) and of seclusion measures on mental health and on the development of psychological disorders in children in the short to medium term

DETAILED DESCRIPTION:
In the context of a viral outbreak and of widespread quarantine measures, a significant increase in psychological disorders, such as stress or fear behaviours, had previously been observed. This distress has been described on adults, but no data have been collected yet for paediatric populations.

After a traumatic event, children and adolescents may present several clinical consequences, the most common being Post-Traumatic Stress Disorder (PTSD). Moreover, PTSD in children and adolescents is often associated with comorbid disorders, such Attention Deficit Hyperactivity Disorder, depression, attachment and anxiety disorders, sleep disturbances and behavior problems.

The aim of this study is to present the methodology of "CoCo 20" : is to assess the impact of the pandemic of coronavirus disease (Covid-19) and of seclusion measures on mental health and on the development of psychological disorders in children in the short to medium term.

The major inclusion criteria are children and adolescents under 18 years of age who have been affected by the Covid 19 pandemic. Three groups were defined: children in group one had a previous history of traumatic events, those in group two had a record of previous psychiatric or psychological disorder with a follow-up treatment and Group three included children without traumatic history nor psychiatric or psychological follow-up treatment. Participants will be assessed at baseline (V0), 1 week after (V1), one month after baseline (V2), one week after the end of the containment (V3) and one month after the end of the containment (V4).

Main analyses comprise analyses of variance and regression analyses of predictors of clinical evolution over time

ELIGIBILITY:
Inclusion Criteria:

* Children affected by the Coronavirus disease 2019 (Covid-19) pandemic;
* Age between 0 and under 18 at the time of inclusion;
* Affiliated with a social security scheme;
* Having a good command of the French language (French);
* Children whose parents have accepted participation in the study (collection of informed consents).

Exclusion Criteria:

* Children and/or young adults with a psychotic disorder or autism spectrum disorder;
* Children and/or young adults with an average intellectual disability (< to 50);
* Person deprived of liberty by judicial or administrative decision1;
* Person subject to a period of exclusion for another search.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Group 1 (PTSD): children with an identified traumatic history; Group 2 (Pathology): children with psychological follow-up treatment for a psychiatric disorder, without traumatic history; Group 3 (Control): children without traumatic experience and without psychiatric or psychological follow-up treatment.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
diagnosis of possible psychological and psychiatric difficulties at baseline | at baseline Day 0
  measure of psychological and psychiatric difficulties in connection with the pandemic and confinement. This will allow a rapid implementation of a course of care adapted and specific to the difficulties presented by each child, by Quantitative and qualitative assessments :

SECONDARY OUTCOMES:
follow up of psychological and psychiatric difficulties at V2 | at one month after baseline
  measure of psychological and psychiatric difficulties in connection with the pandemic and confinement. This will allow a rapid implementation of a course of care adapted and specific to the difficulties presented by each child, by Quantitative and qualitative assessments
follow up of psychological and psychiatric difficulties at V3 | at one week after the end of the containment
  measure of psychological and psychiatric difficulties in connection with the pandemic and confinement. This will allow a rapid implementation of a course of care adapted and specific to the difficulties presented by each child, by Quantitative and qualitative assessments
follow up of psychological and psychiatric difficulties at V4 | at one month after the end of the containment
  measure of psychological and psychiatric difficulties in connection with the pandemic and confinement. This will allow a rapid implementation of a course of care adapted and specific to the difficulties presented by each child, by Quantitative and qualitative assessments
impact of traumatic history prior to confinement | at one week after baseline and at one month after the end of the containment
  measure by Post-Traumatic Stress Disorder (PTSD) scale: The frequency and intensity of PTSD symptoms will be assessed using the Young Child PTSD Checklist (YCP) for children aged 3 months to 6 years and 11 months; or the Child PTSD checklist (CPC) for children aged 7 years to 17 years and 11 months ; or with the Post-Traumatic Stress Disorder ( PTSD) checklist 5 (PCL 5 ) for adults
impact of other previous psychiatric disorders | at one month after baseline and at one month after the end of the containment
  measure by Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS): This is a semi-directed interview for children over the age of 7. It is done by interviewing the parent and the child. The interview covers both current issues.
parental reaction | at one week after baseline and at one week after the end of the containment
  measure by Parenting stress index-short form (PSI-SF) that measures the extent of parental stress, as well as stress in the relationship between parent and child, and parents' difficulties in the day-to-day management of children.

CONTACTS AND LOCATIONS:
Overall Officials: Florence Gittard-Askenazy, Pr, Study Director — Hôpitaux Pédiatriques de Nice CHU-LENVAL
Locations (1):
- Hôpitaux Pédiatriques de Nice CHU-Lenval, Nice, France

REFERENCES:
- [Derived] Gindt M, Fernandez A, Richez A, Nachon O, Battista M, Askenazy F. CoCo20 protocol: a pilot longitudinal follow-up study about the psychiatric outcomes in a paediatric population and their families during and after the stay-at-home related to coronavirus pandemic (COVID-19). BMJ Open. 2021 Apr 8;11(4):e044667. doi: 10.1136/bmjopen-2020-044667. PMID 34270445